CLINICAL TRIAL: NCT04916106
Title: Effect of Transcutaneous Electroacupuncture on Patients With Functional Abdominal Bloating/Distension
Brief Title: Effect of Transcutaneous Electroacupuncture on Functional Abdominal Bloating/Distension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018079; S2020-YF-YBSF-0237 (Other: Shaanxi Provincial Health and Family Planning Commission)
Record Dates: First submitted 2021-05-20; First posted 2021-06-07 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-06

CONDITIONS: Functional Abdominal Bloating/Distension
Keywords: Functional Bloating/Distension; Transcutaneous electrical acupoint stimulation
MeSH Terms: conditions — Dilatation, Pathologic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One parameter TEA group for 4 weeks (Experimental): Choose two acupoints,give 25Hz electrical stimulation for 4 weeks.
  Interventions: Device: Transcutaneous Electroacupuncture
- Another parameter TEA group for 4 weeks (Experimental): Choose two acupoints,give 100 Hz electrical stimulation for 4weeks.
  Interventions: Device: Transcutaneous Electroacupuncture
- Sham-TEA group for 2 weeks, and the random TEA for the next 2 weeks. (Experimental): Choose two non-acupoints，give 25Hz and 100Hz electroacupuncture stimulation respectively for the first 2 weeks. Then give supplement TEA treatment as described above for the next 2 weeks.
  Interventions: Device: Transcutaneous Electroacupuncture

INTERVENTIONS:
Device: Transcutaneous Electroacupuncture — give diffrent parameter TEA treatment for 4 weeks.

SUMMARY:
Functional abdominal bloating/distension (FAB/D) is a common functional bowel disorder that lacks effective treatment options. Transcutaneous electroacupuncture (TEA) as a new therapeutic method has great effect on functional gastrointestinal diseases such as functional dyspepsia and functional constipation. Research on TEA for FAB/D has not yet been explored.

DETAILED DESCRIPTION:
Functional abdominal bloating/distension (FAB/D) is a common functional bowel disorder that lacks effective treatment options. Rome IV was introduced in 2016. Studies have shown that bloating may affect about 30% general population and 96% of patients with functional gastrointestinal disorders (FGID).Transcutaneous electroacupuncture (TEA) as a new therapeutic method has great effect on functional gastrointestinal diseases such as functional dyspepsia and functional constipation. Research on TEA for FAB/D has not yet been explored. Thirty patients who fulfilled the Rome IV diagnostic criteria of FAB/D in the department of the second affiliated hospital of Xi'an jiaotong University.Inclusion criteria included: Symptoms of recurrent abdominal fullness, pressure, or a sensation of trapped gas (bloating), and/or measurable (objective) increase in abdominal girth (distention) more than 6 month；the main symptoms appeared in the past 3 months；Not taking related drugs; aged 18-65 years old；From January 2020 to December 2021; Sign informed consent. All patients were randomly assigned to 3 groups and received TEA at Zusanli (ST36) and Neiguan (PC6) with 3 diffrent parameter for 4weeks. The symptom severity score, abdominal girth, electrogastrogram (ECG) and orocecal transit time (OCTT) ,heart rate variability (HRV) ,rectal sensitivity and intestinal flora were recorded at baseline and after 2-week treatment, respectively. The symptom severity score was repeated at baseline and after 4-week treatment. Through the comparison of the index before and after TEA treatment to identify optimal stimulation parameters and explore its possible mechanism. The study was proved by the medical ethics committee of the Second Affiliated Hospital of Xi'an jiaotong University.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Functional bloating/distension with Rome IV;
2. Aged 18-65 years old；

Exclusion Criteria:

1. Have taken drugs that may affect gastrointestinal motility in the past week;
2. Have taken antibiotics and probiotics in the past month;
3. The history of gastrointestinal surgery;
4. Helicobacter pylori is not cleared；
5. Pregnant and breastfeeding women;
6. Skin allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Symptom improvement rate | after 1 month TEA treatment
  the symptom severity score with VAS and abdominal girth measurements
The percentage of the normal gastric slow waves in electrogastrograph | after 1 month TEA treatment
  The percentage of the normal gastric slow waves in fasting 、fed states and the post-preprandial EGG power ratio
Orocecal ransit time | after 1-month TEA treatment
  the lactulose hydrogen breath test was used to evaluate the intestinal transit time and observe the presence or absence of excessive small intestinal bacteria
Heart rate variability（HRV） | after 1-month TEA treatment
  Assessment of autonomic function with heart rate variability
Flora structure | after 1-month TEA treatment
  an Illumina MiSeq Platform was used to sequence 16S ribosomal RNA (rRNA) gene of the total bacteria in fecal samples.
Rectal sensitivity | after 1-month TEA treatment
  Rectal threshold for gas and defecation
Plasma gastrointestinal peptide level | after 1-month TEA treatment
  CCK、SP、NPY、CGRP、Motilin

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China